CLINICAL TRIAL: NCT05402176
Title: Silicosis - Harnessing New Ideas to Conquer the Re-emergence of an Ancient Lung Disease: The SHIELD Whole Lung Lavage Study
Brief Title: The SHIELD Whole Lung Lavage Study
Acronym: SHIELD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: SHIELD WLL
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Silicosis
MeSH Terms: conditions — Silicosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Biomarkers (blood ACE and ferritin) and WLL effluent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Whole Lung Lavage — Whole Lung Lavage (WLL) is performed as standard of care. Outcome following WLL is observed.

SUMMARY:
An observational cohort study that will assess the efficacy of Whole Lung Lavage in workers with silicosis or silica-induced bronchitis.

DETAILED DESCRIPTION:
BACKGROUND: Silicosis is a fatal lung disease caused by inhaling silica particles. Australia is currently facing an epidemic with hundreds of young workers having contracted silicosis from machining engineered stone.

AIMS: To determine the effectiveness and safety of Whole Lung Lavage (WLL) in workers with silicosis due to significant engineered stone exposure.

DESIGN: Participants (30) with silicosis or silica-induced bronchitis who are scheduled to undergo WLL as part of their normal care will be enrolled. They will undergo the following interventions pre and 3 months post WLL, some of which would have been carried out as part of routine standard care:

1. Complex pulmonary function tests (PFTs) - standard care
2. HRCT scan (if not within 6 months of WLL) - standard care
3. Blood tests
4. Cardiopulmonary exercise testing
5. Forced oscillatory technique
6. XV Lung Ventilation Analysis
7. Questionnaires (K-BILD and LCQ)

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged >=18 years and scheduled for WLL at the study site as part of routine clinical care
* History of exposure to respirable crystalline silica (RCS) while working in an at-risk industry (e.g. stonemasonry, construction, tunnelling, concreting, mining)
* Elimination of workplace exposure to RCS for a minimum of 6 months
* Ground glass nodularity > extent of solid nodularity on HRCT, as judged by investigator or evidence of silica-induced bronchitis
* Evidence of disease progression within the past 2 years, defined as any of

  * a relative decline in the FVC or FEV1 of at least 5% of the predicted value,
  * worsening of respiratory symptoms
  * increased extent of silicosis on high-resolution CT scan
* Able to understand and sign a written informed consent form (or legally authorised representative)

Exclusion Criteria:

* Ongoing workplace exposure to RCS or removal of workplace exposure of less than 6 months
* Progressive massive fibrosis, defined as areas of confluent fibrosis with diameter > 10mm on HRCT.
* FEV1 or FVC < 50% predicted
* DLCO <50% predicted
* Contraindication to WLL, as judged by the investigator
* Actively or imminently listed for lung transplantation
* Females with a positive pregnancy test at screening or currently breastfeeding
* Any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next 24 months
* Any condition other than silicosis that, in the opinion of the investigator, is likely to result in the death of the participant within the next 24 months
* Significantly impaired cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respirable crystalline silica (RCS) exposed workers with silicosis or silica induced bronchitis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome for evaluating WLL will be change in dual blind read CT ICOERD score from baseline to 3 months post WLL. | 3 months
  Change in absolute dual-read CT ICOERD score at 3 months post-WLL. Data collected will be evaluated by a central reader blinded to treatment assignment. Baseline characteristics will be summarised for each group. Differences between group mean changes in CT ICOERD scores from baseline to 3 months will be tested using an independent sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chambers, Principal Investigator — The Prince Charles Hospital
Locations (4):
- Australia (4):
  - The Royal Prince Alfred Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - The Austin Hospital, Melbourne, Victoria